CLINICAL TRIAL: NCT06417294
Title: Effects of a 3D-Printed Port-A Catheter Model Training Course for Patient Discharge Instruction
Brief Title: Effects of a 3D-Printed Port-A Catheter Model Training Course
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH112278
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Patient Satisfaction; Cancer
Keywords: 3D printed model; port-a catheter; discharge education
MeSH Terms: conditions — Patient Satisfaction; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D model group (Experimental): Received a explanation combined with 3D printed model
  Interventions: Other: 3D health education model
- traditional education group (Active Comparator): Received a regular education
  Interventions: Other: traditional education

INTERVENTIONS:
Other: 3D health education model — explanation combined with 3D printed health education model
  Arms: 3D model group
Other: traditional education — Regular education
  Arms: traditional education group

SUMMARY:
The aim of this study is to develop a highly realistic 3D-printed Port-A catheter upper body model to improve the knowledge and self-care skills of patients and primary caregivers regarding Port-A catheter placement through patient education.

DETAILED DESCRIPTION:
Background： Cancer patients often require long-term administration of chemotherapy drugs, nutritional supplementation, and blood transfusions. During these treatments, an implantable central venous access (port-a catheter) is often utilized to avoid the inconvenience of repeated needle insertions for treatment and to minimize the risk of medication leakage. Port-A catheters are considered a safer clinical measure. However, poor care and maintenance of the catheter can lead to complications such as infection, catheter damage, and leakage, which can even result in death. The study aims to assess the impact of patient discharge education on their knowledge and satisfaction regarding catheter care.

Methods： This study focuses on patient education and evaluating its effectiveness. It employs a prospective randomized controlled trial with a cross-sectional design and parallel groups. The participants are divided into the 3D model group (experimental group) and the conventional education group (control group). A total of 120 subjects from the hematology-oncology ward are included in the study. The participants are randomly assigned to either the experimental group (60 participants) or the control group (60 participants) based on the month of admission, following a cluster randomization approach.

Effect： The investigator anticipate that the use of a 3D-printed upper body Port-A catheter model will yield better results in patient discharge education.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hematology and oncology ward of Fu Jen Catholic University Hospital
* Have Chinese communication skills

Exclusion Criteria:

* Refused to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient education effectiveness questionnaire | immediately after the intervention
  higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No